CLINICAL TRIAL: NCT04743037
Title: Feasibility of Mobile Self-Management Intervention for Mild Stroke
Brief Title: Interactive Self-Management Augmented by Rehabilitation Technologies
Acronym: iSMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202004137
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Occupational Therapy; Epidemiology; Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): The 15 attentional control group stroke survivors will receive phone calls over the 12-week intervention checking in with them on how they are doing in their everyday life. They will also receive stroke education materials, but they will not receive the same iSMART intervention as the intervention group.
- iSMART (Experimental): The 15 iSMART participants will engage in video conference sessions between the pre and post visits. A health coach will collaboratively work with the participant to practice treatment strategies and set goals in weekly individual sections. In addition, all participants will engage in weekly group sessions with a health coach in order to learn and practice specific self-management skills and strategies in a group context. In addition, iSMART entails using an interactive SMS to provide ongoing support and self-monitoring of behavior change goals. The SMS is programmed to "touch" participants daily; the SMS system prompts participants to report their daily activities and progress in achieving goals via "check-in" messages and sends immediate, tailored feedback about their progress. If a participant is making progress toward their goal, the SMS system will suggest a change to the participant's goal between visits.
  Interventions: Behavioral: iSMART

INTERVENTIONS:
Behavioral: iSMART — This patient-centered and participation-focused self-management intervention will help individuals develop strategies to manage chronic conditions and support their full participation in meaningful life activities.
  Arms: iSMART

SUMMARY:
Background: Stroke is a leading cause of long-term disability in the US. Mild stroke comprises half of stroke hospital admissions, but most people with mild stroke receive no rehabilitation services. Mild stroke is often the manifestation of uncontrolled chronic conditions (e.g. hypertension, diabetes), and people with mild stroke also experience ongoing chronic symptoms (e.g. depression, fatigue) that may impact their daily activities. An inability to manage chronic conditions and symptoms may lead to decreased participation in pre-stroke roles and activities, which may increase the chance of sustaining a second stroke. An effective intervention to manage chronic conditions and support participation is self-management. A meta-review of 13 systematic reviews demonstrated that self-management interventions significantly improve stroke survivors' daily activities, independence, and mortality. National research agendas from the Department of Health and Human Services (HHS) and Institute of Medicine (IOM) include self-management as one key goal of a strategic framework, aligning with the AOTF Research Priorities, for promoting (1) health behaviors to prevent and manage chronic conditions. Our preliminary studies indicate that mobile health (mHealth), defined as the delivery of healthcare services via mobile devices, can be used to precisely monitor participation in daily activities and mood and is acceptable in stroke survivors. Our meta-analysis indicates that digital self-management interventions are more effective in improving depression, fatigue, anxiety, and self-efficacy in people with neurologic disorders in comparison to non-digital self-management interventions. These studies support the AOTF Research Priorities that include (2) use of technology to support home and community activities, and (3) emotional influences.

Objectives: The investigators will harness mHealth technology for a self-management program. Our intervention is a mobile phone intervention called iOTA, which builds on extensive work by my mHealth mentor and colleagues in health behavior research. The investigators will use a formal implementation science framework to adapt and test the iOTA intervention. The investigators will cohere an adaptation framework by soliciting stakeholder input to adapt the iOTA from Improving Participation after Stroke Self-Management (IPASS), an evidence-based intervention that targets self-management of chronic conditions and increased community participation in stroke survivors.

Methods: The investigators will use a two-step approach, including a rigorous treatment adaptation and a Phase I feasibility trial. Our first step is to adapt the intervention with input from all relevant stakeholder levels. Our second step is to use a pre-post, non-randomized study design to test the adapted iOTA. Ten community-dwelling people with mild stroke will participate in the iOTA for 3 months. The iOTA incorporates daily short message service (SMS) text messages to supplement monthly in-person health coaching and weekly videoconference sessions. The investigators will include an occupational therapist (OT) as a health coach to teach individuals to incorporate self-management strategies into their daily routines to support participation in meaningful activities.

Expected Outcome: This mHealth treatment development study will increase the reach and access of IPASS-a patient-centered, participation-focused self-management program for stroke survivors. The iOTA created will not only maximize our potential for the future randomized controlled trial (RCT) but also lay the groundwork for future funding mechanisms.

DETAILED DESCRIPTION:
In this study, the investigators will take 30 stroke survivors and have them participate in a 3-month study consisting of screening, assessments, goal setting, health coaching, EMA surveys, and feedback on how to improve the study for a future expanded study.

After the research team consents and enrolls participants, participants will be randomized and complete screening, assessment, and training on the video conferencing system, training on the Status/Post and SMS. The screening measures and assessments that will be performed are: Participation Strategies Self-Efficacy Scale, PROMIS Self Efficancy, Stroke Impact Scale, Activity Card Sort, Reintegration to Normal Living Index, PHQ-9, PROMIS 29+2, Light House Test, Boston Naming Test, and Short Blessed Test form are all assessments that will be performed online through REDCap via a secure link over the phone or email. The last three tests are screening instruments. The investigators can perform all assessments online through REDCap via a secure link over the phone or email. All data collected will be directly entered into REDCap. Participants will receive an iPod touch if they do not have an iPhone which will be mailed to them to use for the next 14 days. Participants will complete the EMA assessment prototype 5x/day for 14 days via the Status/post-application. Goals will also be set that the participant would like to achieve. If participants do not have a phone or mobile device capable of using the video conferencing system and SMS, the investigators will mail them an iPad to use for the study duration.

The 15 MyIPASS participants will engage in video conference sessions between the pre and post visits. A health coach will collaboratively work with the participant to practice treatment strategies and set goals in weekly individual sections. In addition, all participants will engage in weekly group sessions with a health coach in order to learn and practice specific self-management skills and strategies in a group context. In addition, MyIPASS entails using an interactive SMS to provide ongoing support and self-monitoring of behavior change goals. The SMS is programmed to "touch" participants daily; the SMS system prompts participants to report their daily activities and progress in achieving goals via "check-in" messages and sends immediate, tailored feedback about their progress. If a participant is making progress toward their goal, the SMS system will suggest a change to the participant's goal between visits.

The 15 attentional control group stroke survivors will receive phone calls over the 12-week intervention checking in with them on how they are doing in their everyday life. They will also receive stroke education materials, but they will not receive the same MyIPASS intervention as the intervention group.

A pre-selected time will be scheduled for the participant to complete their post-assessments, and complete an interview after the 12 weeks via the phone. The assessments will be administered the same as they were in the pre-test, given a link over the phone or email to a secure RedCap site which will include the following assessments: Client Satisfaction Questionnaire (CSQ), Healing Encounters & Attitudes Lists - Patient-Provider Connection (HEAL-PPC), PROMIS Self Efficancy, Stroke Impact Scale, Activity Card Sort, Reintegration to Normal Living Index, PHQ-9, PROMIS 29+2, Acceptability of Implementation Measure (AIM), Appropriateness of Implementation Measure (IAM), and Feasibility of Implementation Measures after the intervention. The investigators will ask them to mail the iPod back to the lab when they are finished with their 14-day surveys with a prepaid envelope. If participants used an iPad, they will return it to the lab via mail in a prepaid envelope.

At the conclusion of the trial, the investigators will ask the 30 stroke survivors, the investigators will conduct the feedback questions during the follow-up phone appointment. All interviews will be facilitated by a moderator. Moderators will be trained with the interview guide and Computer Usage Questionnaire. Sessions will be audio/video recorded to allow for transcription and analysis. Participants may share as much as they would like or feel comfortable.

Data from participants will be collected from screening measures, assessments, and the SMS prototype. Please refer to the attachment for knowing what coded data will be extracted from the SMS dashboard. During the data collection process, members of the research team may photograph the participant doing a variety of tasks if given permission.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhagic stroke (NIHSS scores ≤13)
* aged ≥18
* English-speaking
* ≥3 months post-stroke
* identified as having ≥1 chronic condition
* mobile phone ownership.

Exclusion Criteria:

* previous neurologic or psychiatric disorder (e.g. dementia or schizophrenia)
* Short Blessed Test score ≥9 (indicating severe cognitive impairment) (Katzman et al., 1983)
* history of functional problems (pre-morbid modified Ranking Scale score ≥2) regardless of prior stroke
* severe aphasia (Boston Naming Test ≤10) (Kaplan, Goodglass, & Weintraub, 2001) or NIH Stroke Scale Aphasia subscale score ≥2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability: Acceptability of Intervention Measure (AIM) | Post-treatment (week 12)
  A 4-item short-form to assess acceptability of an intervention's implementation (Weiner et al., 2017). High acceptability is defined as the score 16 or higher out of 20 on the AIM.
Appropriateness: Intervention Appropriateness Measure (IAM) | Post-treatment (week 12)
  A 4-item short-form to assess appropriateness of an intervention's implementation (Weiner et al., 2017). High appropriateness is defined as the score 16 or higher out of 20 on the IAM.
Feasibility: Feasibility of Intervention Measure (FIM) | Post-treatment (week 12)
  A 4-item short-form to assess feasibility of an intervention's implementation (Weiner et al., 2017). High feasibility is defined as the score 16 or higher out of 20 on the FIM.
Satisfaction: Client Satisfaction Questionnaire | Post-treatment (week 12)
  An 8-item measure to assess the extent of satisfaction with services and met needs (Attkisson & Greenfield, 2004). High acceptability is defined as the score 24 or higher out of 32 on the Client Satisfaction Questionnaire.
Participation Self-Efficacy: Participation Strategies Self-Efficacy Scale | Pre-treatment (week 0) and Post-treatment (week 12
  A 35-item measure to assess the self-efficacy in managing home, work, community participation; communication; & advocating resources (D. Lee, Fogg, Baum, Wolf, & Hammel, 2018). Pre- and post-treatment change score is used to indicate the magnitude change of this construct after intervention. Cohen's d effect size of change >.20 to indicate a meaningful change.
General Self-Efficacy: PROMIS-Self-Efficacy Short Forms | Pre-treatment (week 0) and Post-treatment (week 12)
  5 short forms to assess self-efficacy for managing: (1) daily activities, (2) medications and treatment, (3) symptoms, (4) emotions, and (5) social interactions. Each form is consisted of 4 items (Gruber-Baldini, Velozo, Romero, & Shulman, 2017). Pre- and post-treatment change score is used to indicate the magnitude change of this construct after intervention. Cohen's d effect size of change >.20 to indicate a meaningful change.

SECONDARY OUTCOMES:
Functioning: Stroke Impact Scale | Pre-treatment (week 0) and Post-treatment (week 12)
  A 59-item self-reported scale to measure 8 domains: strength, hand function, ADLs, mobility, communication, emotion, cognition, and participation (Duncan, Bode, Lai, & Perera, 2003). Pre- and post-treatment change score is used to indicate the magnitude change of this construct after intervention. Cohen's d effect size of change >.20 to indicate a meaningful change.
Activity: Activity Card Sort | Pre-treatment (week 0) and Post-treatment (week 12)
  A 89-item measure to assess the engagement in social, instrumental, & leisure activities (C. M. Baum & Edwards, 2001). Pre- and post-treatment change score is used to indicate the magnitude change of this construct after intervention. Cohen's d effect size of change >.20 to indicate a meaningful change.
Participation: Reintegration to Normal Living Index | Pre-treatment (week 0) and Post-treatment (week 12)
  An 11-item measure to assess the extent of integration into normal activities after illness (Bourget, Deblock-Bellamy, Blanchette, & Batcho, 2018). Pre- and post-treatment change score is used to indicate the magnitude change of this construct after intervention. Cohen's d effect size of change >.20 to indicate a meaningful change.
Quality of Life: PROMIS® 29+2 Profile v2.1 (PROPr) | Pre-treatment (week 0) and Post-treatment (week 12)
  PROPr is used to calculate a preference score. This preference-based score is estimated based on multiple health domains (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognitive abilities), which provides a single summary score for overall health that can be used in comparisons across groups, treatment options in decision-making and cost-effectiveness analyses. We will also use this instrument throughout individual coaching sessions to guide the participant to identify the key problem area for self-management (Dewitt et al., 2018). Pre- and post-treatment change score is used to indicate the magnitude change of this construct after intervention. Cohen's d effect size of change >.20 to indicate a meaningful change.
Non-specific treatment factors: Healing Encounters & Attitudes Lists | Course of Study 12 weeks
  : Measuring nonspecific factors in treatment, including: (1) patient-provider connection (PPC), (2) healthcare environment (HCE), (3) treatment expectancy (TE), (4) positive outlook, and (5) spirituality (Greco et al., 2016)

CONTACTS AND LOCATIONS:
Overall Officials: Wing Wong, PhD, Principal Investigator — Washington University OT
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] Li Z, Lei Y, Bui Q, DePaul O, Nicol GE, Mohr DC, Lee SI, Fong MWM, Metts CL, Tomazin SE, Wong AWK. A Digital Intervention to Promote Self-Management Self-Efficacy Among Community-Dwelling Individuals With Stroke: Pilot Randomized Controlled Trial. JMIR Rehabil Assist Technol. 2024 Feb 19;11:e50863. doi: 10.2196/50863. PMID 38373029